CLINICAL TRIAL: NCT05275907
Title: Pilot Study to Assess Blockade of Calcium Channels and Sodium Chloride Cotransporters for Physiologic Abnormalities in Liver Transplant Associated Hypertension
Brief Title: Mechanism of Hypertension Treatments in Liver Transplant Recipients (BLOCK LTR-HTN)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Screened participants did not meet inclusion criteria prior to study completion date
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Society for Transplantation (Unknown)
Responsible Party: Principal Investigator, Dempsey Hughes, Assistant Professor of Medicine-Gastroenterology & Hepatology, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: STU00215781; 1R56HL155093-01 (NIH)
Record Dates: First submitted 2021-11-17; First posted 2022-03-11 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: High Blood Pressure; Liver Transplant; Renal Function Abnormal
Keywords: liver transplant; hypertension; cardiac function; kidney function; treatment
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A first, then B (Active Comparator): 6 weeks of drug A followed by a 2-week washout period completed with 6 weeks of drug B
  Interventions: Drug: Amlodipine Besylate; Drug: Chlorthalidone
- B first, then A (Active Comparator): 6 weeks of drug B followed by a 2-week washout period completed with 6 weeks of drug A
  Interventions: Drug: Amlodipine Besylate; Drug: Chlorthalidone

INTERVENTIONS:
Drug: Amlodipine Besylate — 10 mg capsule once daily for 6 weeks
Drug: Chlorthalidone — 25mg capsule once daily for 6 weeks

SUMMARY:
Liver transplantation is a high risk, high-cost intervention that extends life in over 8,000 patients in the US each year. Of those that receive transplants, 1 in 3 will have a complication related to their heart after transplant. Research has been done to attempt to reduce the risk of these complications from occurring. High blood pressure, otherwise known as "hypertension," is an important risk factor for heart complications. Hypertension is found in 92% of liver transplant recipients within 6 years of their procedure. However, using data from our transplant patients at Northwestern we recently showed that having a normal blood pressure in the first year following liver transplant lowered the risk of heart complications and the risk of death by over half. However, there are no studies investigating the best medications to lower blood pressure in liver transplant recipients.

There are several types of medications that can be used to treat high blood pressure. Currently, most transplant providers use a class of medications called calcium channel blockers as the first medications for hypertension in liver transplant patients. However, there is little data to support this recommendation. There is some new evidence suggesting that another class of medications, called thiazide-like diuretics, might be beneficial to lower blood pressure in liver transplant recipients. The current study will use two different medications: the calcium channel blocker called amlodipine besylate (at dose of 10mg) and the thiazide-like diuretic known as chlorthalidone (25mg). Both medications are taken once per day by mouth and are FDA approved for the treatment of high blood pressure in the general population.

The main purpose of this study is to determine how well these two medications lower blood pressure and how they may improve markers of heart function and kidney function in liver transplant recipients. The long-term goal of this research is to improve heart outcomes in those that have undergone liver transplant by addressing risk factors that can be modified, including blood pressure. This study will help determine the size of the needed group for further studies to ensure proper investigation of which of these two medications may most benefit liver transplant patients.

DETAILED DESCRIPTION:
The study will involve a randomized crossover trial of two medications: amlodipine besylate 10mg and chlorthalidone 25mg daily by mouth. Amlodipine was selected as the dihydropyridine calcium channel blocker (CCB) due to extensive trial evidence demonstrating its efficacy in hypertension (HTN) in the general population and established safety and efficacy for calcineurin inhibitor (CNI)-induce HTN in kidney transplant recipients. Chlorthalidone was chosen amongst other thiazides due to its favorable safety profile, superior effectiveness in reducing cardiovascular events (CVEs) in the general population, stronger reduction in central pressure, and prior evidence of efficacy in kidney transplant recipients with CNI-induced HTN. Dosing for either medication was determined based on the median and maximum recommended doses for each medication when used for the treatment of stage II HTN BP ≥140/≥90 and previous trial evidence demonstrating similar blood pressure-lowering effects of amlodipine and chlorthalidone at these doses. We recognize that several prior studies have used a starting dose of chlorthalidone 12.5mg; however, this dose is no longer available in the U.S. and tablets are not scored to allow for accurate trial dosing. We specifically selected a relatively short duration of follow up (six weeks per intervention) due to several factors, including 1) the time to peak hemodynamic effects and durations of action of the trial interventions, balanced with 2) optimizing adherence to the study protocols to be able to measure key mechanistic factors, and 3) minimizing dropout. Given the well-described half-life elimination of the two medications, we do not anticipate issues with crossover effects in the second phase outcome assessments occurring six weeks following the washout period. Nonetheless, exploratory analyses will account for potential period or crossover effects using mixed effects models.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant alone recipient
* At least 90 days from transplant
* Average daytime systolic blood pressure (SBP)>140mmHG with 24h ambulatory blood pressure monitoring. Patients will be enrolled in 24h ambulatory blood pressure monitoring (ABPM) if they have hypertension (HTN) defined by diagnostic codes, treatment with antihypertensive medications for ≥ 2 months, and a history of office blood pressure readings ≥140/90 mmHg at two separate office visits.
* Stable antihypertensive medical therapy (e.g., no change in current antihypertensive medications within 30d of screening)
* No acute cellular rejection within 30d of screening

Exclusion Criteria:

* Contraindication to withholding calcium channel blockers (CCB) or beta-blocker (e.g., atrial fibrillation/flutter)
* Treatment with other diuretics that cannot be held
* Acute coronary syndrome or revascularization within 60d
* Serum potassium < 3.5 mEq/L
* Serum sodium < 135 mg/dL
* Allergy to sulfa drugs
* Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m2 or on dialysis
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Change in central aortic pressure at 6 weeks of therapy compared to baseline values | Endpoints will be measured before the first dose of either amlodipine or chlorthalidone and at the end of each six-week double-blinded treatment period
  Carotid-femoral pulse wave velocity (PWV), the gold standard measure of large artery stiffness, will be measured using a SphygmoCor XCEL device (Atcor Medical).

SECONDARY OUTCOMES:
Number of patients with improvement in diastolic function (E/e' ratio) | Endpoints will be measured before the first dose of either amlodipine or chlorthalidone and at the end of each six-week double-blinded treatment period
  We will perform comprehensive echo to assess diastolic function using E/e' ratio on all participants using a GE Vivid T8 ultrasound machine and a systematic echo protocol.
Number of patients with improvement in systolic function (absolute global longitudinal strain, %) | Endpoints will be measured before the first dose of either amlodipine or chlorthalidone and at the end of each six-week double-blinded treatment period
  We will perform comprehensive echo to assess systolic function using absolute global longitudinal strain (%) on all participants using a GE Vivid T8 ultrasound machine and a systematic echo protocol.
Change in Blood pressure | Endpoints will be measured before the first dose of either amlodipine or chlorthalidone and at the end of each six-week double-blinded treatment period
  24-hour ambulatory blood pressure (BP) monitoring will be performed in addition to office BP to determine Mean home systolic and diastolic BP, office systolic and diastolic BP and nocturnal BP readings
Change in Renal function | Endpoints will be measured before the first dose of either amlodipine or chlorthalidone and at the end of each six-week double-blinded treatment period
  Renal function will be primarily assessed by 24-hour creatinine clearance which is the most accurate measure of GFR after liver transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Dempsey Hughes, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification
Supporting Information: Study Protocol
Time Frame: Following publication with no end date.
Access Criteria: Any purpose.

REFERENCES:
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2018 May 15;71(19):e127-e248. doi: 10.1016/j.jacc.2017.11.006. Epub 2017 Nov 13. No abstract available. PMID 29146535
- [Background] ALLHAT Officers and Coordinators for the ALLHAT Collaborative Research Group. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Major outcomes in high-risk hypertensive patients randomized to angiotensin-converting enzyme inhibitor or calcium channel blocker vs diuretic: The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). JAMA. 2002 Dec 18;288(23):2981-97. doi: 10.1001/jama.288.23.2981. PMID 12479763
- [Background] Wright JT Jr, Dunn JK, Cutler JA, Davis BR, Cushman WC, Ford CE, Haywood LJ, Leenen FH, Margolis KL, Papademetriou V, Probstfield JL, Whelton PK, Habib GB; ALLHAT Collaborative Research Group. Outcomes in hypertensive black and nonblack patients treated with chlorthalidone, amlodipine, and lisinopril. JAMA. 2005 Apr 6;293(13):1595-608. doi: 10.1001/jama.293.13.1595. PMID 15811979
- [Background] Dahlof B, Sever PS, Poulter NR, Wedel H, Beevers DG, Caulfield M, Collins R, Kjeldsen SE, Kristinsson A, McInnes GT, Mehlsen J, Nieminen M, O'Brien E, Ostergren J; ASCOT Investigators. Prevention of cardiovascular events with an antihypertensive regimen of amlodipine adding perindopril as required versus atenolol adding bendroflumethiazide as required, in the Anglo-Scandinavian Cardiac Outcomes Trial-Blood Pressure Lowering Arm (ASCOT-BPLA): a multicentre randomised controlled trial. Lancet. 2005 Sep 10-16;366(9489):895-906. doi: 10.1016/S0140-6736(05)67185-1. PMID 16154016
- [Background] Luscher TF, Yang Z, Kiowski W, Linder L, Dohi Y, Diederich D. Endothelin-induced vasoconstriction and calcium antagonists. J Hum Hypertens. 1992 Dec;6 Suppl 2:S3-8. PMID 1289511
- [Background] Neal DA, Brown MJ, Wilkinson IB, Byrne CD, Alexander GJ. Hemodynamic effects of amlodipine, bisoprolol, and lisinopril in hypertensive patients after liver transplantation. Transplantation. 2004 Mar 15;77(5):748-50. doi: 10.1097/01.tp.0000116418.78963.dc. PMID 15021839
- [Background] Levitsky J, O'Leary JG, Asrani S, Sharma P, Fung J, Wiseman A, Niemann CU. Protecting the Kidney in Liver Transplant Recipients: Practice-Based Recommendations From the American Society of Transplantation Liver and Intestine Community of Practice. Am J Transplant. 2016 Sep;16(9):2532-44. doi: 10.1111/ajt.13765. Epub 2016 Apr 22. PMID 26932352
- [Background] Moes AD, Hesselink DA, van den Meiracker AH, Zietse R, Hoorn EJ. Chlorthalidone Versus Amlodipine for Hypertension in Kidney Transplant Recipients Treated With Tacrolimus: A Randomized Crossover Trial. Am J Kidney Dis. 2017 Jun;69(6):796-804. doi: 10.1053/j.ajkd.2016.12.017. Epub 2017 Mar 1. PMID 28259499
- [Background] Olde Engberink RH, Frenkel WJ, van den Bogaard B, Brewster LM, Vogt L, van den Born BJ. Effects of thiazide-type and thiazide-like diuretics on cardiovascular events and mortality: systematic review and meta-analysis. Hypertension. 2015 May;65(5):1033-40. doi: 10.1161/HYPERTENSIONAHA.114.05122. Epub 2015 Mar 2. PMID 25733241
- [Background] Kwon BJ, Jang SW, Choi KY, Kim DB, Cho EJ, Ihm SH, Youn HJ, Kim JH. Comparison of the efficacy between hydrochlorothiazide and chlorthalidone on central aortic pressure when added on to candesartan in treatment-naive patients of hypertension. Hypertens Res. 2013 Jan;36(1):79-84. doi: 10.1038/hr.2012.143. Epub 2012 Oct 4. PMID 23034468
- [Background] Pareek A, Messerli FH, Saravia G, Mehta RT. Interamerican Society of Cardiology (IASC) position statement: Chlorthalidone vs. thiazide-type diuretics. Int J Cardiol Hypertens. 2020 Sep 19;7:100054. doi: 10.1016/j.ijchy.2020.100054. eCollection 2020 Dec. PMID 33447776